CLINICAL TRIAL: NCT00619671
Title: Phase 1-2 Pilot Study of Rituximab (Rituxan) in Refractory Myasthenia Gravis.
Brief Title: A Pilot Trial of Rituxan in Refractory Myasthenia Gravis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Dr. Rup Tandan, M.D., F.R.C.P., Professor, University of Vermont
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RituxanMGPilot; BB-IND# 11403; Genentech #U2444S; UVM CHRMS #04-086
Record Dates: First submitted 2008-01-14; First posted 2008-02-21 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Refractory Myasthenia Gravis
Keywords: Rituxan; Rituximab; Myasthenia Gravis; MG
MeSH Terms: conditions — Myasthenia Gravis | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Rituximab (Rituxan) — Four weekly IV infusions of Rituxan with dosage individually calculated per subject.
  Other Names: Rituxan; Rituximab; MabThera

SUMMARY:
Myasthenia gravis is a disease that happens because the immune system attacks the nervous system. The damage is caused by antibodies produced by B lymphocytes. These antibodies damage a special part of the muscle that helps transmit impulses from nerves to muscles to allow muscles to work properly. This damage results in symptoms of myasthenia gravis. Participants are being asked to participate in this research study because their myasthenia gravis has either failed to respond to treatments commonly used in the disease, or they have had bad side-effects from such treatments.

This is a research study of a drug called Rituximab. Rituximab, also called Rituxan, is a mouse antibody that has been changed to make it similar to a human antibody. Antibodies are proteins that can protect the body from foreign invaders, such as bacteria and viruses, by binding to substances called antigens. Rituxan works by binding to a protein, called the CD20 protein. Rituxan helps to destroy white blood cells that produce antibodies in the body, called B-lymphocytes. It is a treatment given through a vein in the participant's arm over a period of approximately 4-6 hours. It has been approved by the Food and Drug Administration (FDA) for use in patients with a form of cancer of the lymph glands called Non-Hodgkin's Lymphoma (NHL). Rituximab is not approved for their myasthenia gravis.

Treatment with Rituximab is being tried in this research study because Rituximab decreases B lymphocytes. There is preliminary evidence that Rituximab helps some patients with chronic and otherwise difficult to treat myasthenia gravis.

DETAILED DESCRIPTION:
Myasthenia gravis (MG) is an immune-mediated disorder of the neuromuscular junction diagnosed on the basis of clinical, electrophysiological and serological features. Cyclosporine as a disease-modifying therapy has been effective in a controlled study; corticosteroids, immunosuppressive agents such as azathioprine and cyclophosphamide, plasmapheresis and intravenous human immune globulin have shown benefit in uncontrolled trials. There are several drawbacks to currently used medical treatments, including serious and debilitating side-effects, prohibitive costs, and the need for continuous or periodical treatment. Almost 20-25% of patients with MG are unresponsive to commonly used therapies, resulting in significant burden and economic loss. Rituximab is a chimeric anti-CD20 monoclonal antibody which produces a substantial reduction in circulating plasma cells (CD19+) and B cells (CD20+) and provides targeted therapy for B-cell lymphomas. Recently, rituximab has been found to be effective in several antibody-mediated autoimmune processes, including immune thrombocytopenia, autoimmune hemolytic anemia, and IgM-related polyneuropathies. There is preliminary evidence in the literature that treatment of MG patients with rituximab is likely to be of benefit. These observations would strongly suggest that rituximab might benefit refractory MG and needs further study.

ELIGIBILITY:
Inclusion Criteria:

Criteria for patient selection will be based upon the recent recommendations for clinical research standards by the Task Force of the Medical Scientific Advisory Board of the Myasthenia Gravis Foundation of America (Jaretzki et al, 2000).

Patients will be included in the trial based upon fulfilling all the criteria given below, except that they will be required to fulfill criterion 3 OR 4:

1. Patients must have a diagnosis of "Definite" MG (Seybold, 1999) as based on clinical, electrophysiological and serological criteria (Appendix 1)
2. Patients must have disease predominantly affecting bulbar or respiratory muscles of moderate or severe degree (Osserman grades 2B, 3 without crisis, or 4 without crisis) (Osserman and Genkins, 1971 and Appendix 2) as listed in Appendix 3, and a Quantitative MG score of <25 (Appendix 7)
3. Patients must have disease refractory to treatment for at least 12 months with prednisone at a dose of 15mg/day and/or immunosuppressive drugs (azathioprine or cyclophosphamide at a dose of 100mg/day or cyclosporine at a dose to produce trough levels of >50), with or without thymectomy and plasmapheresis/IVIG alone or in combination with above drugs at intervals of no more than once every 3 weeks, OR
4. Patients must have experienced intolerance or unacceptable side-effects following treatment with corticosteroids, immunosuppressive drugs (azathioprine, cyclophosphamide or cyclosporine), plasmapheresis or IVIG
5. Patients must be between 18 years and 80 years old
6. Patients must have adequate organ function / laboratory parameters as measured by the following criteria (values should be obtained within 2 weeks prior to enrollment):

   * Documented CD20 + cells
   * Absolute neutrophil count: >2000/mm3
   * Platelets: >100,000/mm3
   * Hemoglobin: >10 gm/dL
   * Adequate renal function as indicated by normal BUN and creatinine levels
   * Adequate liver function, as indicated by AST and ALT <2x Upper Limit of normal.
   * Normal serum electrolytes
7. Men and women of reproductive potential must agree to use an acceptable method of birth control during treatment and for one year after completion of treatment
8. Written informed consent.

Exclusion Criteria:

Patients will be excluded from the trial based on the following criteria:

1. Myasthenic crisis with a forced vital capacity (FVC) of <30% predicted, irrespective of need for respiratory support, or severe bulbar involvement (Appendix 3)
2. Patients requiring maintenance plasmapheresis or IVIG infusions at intervals of less than once every three weeks
3. Patients requiring respiratory support with invasive or non-invasive ventilation
4. Severe, uncontrolled or untreated concomitant cardiac (New York Heart Classification III or IV disease), hepatic, pulmonary, renal, hematologic or psychiatric disease
5. Toxicity grade 2 or more prior to treatment with rituximab in patients who failed prior treatments
6. Patients unwilling to attend for follow-up visits according to the study design
7. Patients will be excluded based on the following criteria:

   * History of HIV disease
   * Active Hepatitis B infection
   * Pregnancy (a serum pregnancy test will be performed for all women of childbearing potential immediately before treatment)
   * Active infection
8. Pregnant or breastfeeding women may not participate due to the lack of information on effects of rituximab on the fetus and developing child
9. Concomitant malignancies or previous malignancies within the last 5 years, with the exception of adequately treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix.
10. No prior monoclonal antibody therapy.
11. History of significant psychiatric disease that will interfere with the consenting procedure, research visits, treatment protocol or evaluation of patients in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2004-04; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
To examine the effects of rituximab on disease activity in MG patients with refractory disease. | Patients will be followed for one year

SECONDARY OUTCOMES:
To determine the safety and tolerability of rituximab in MG patients with refractory disease. | Patients will be followed for one year

CONTACTS AND LOCATIONS:
Overall Officials: Rup Tandan, MD, FRCP, Principal Investigator — University of Vermont Department of Neurology
Locations (2):
- United States (2):
  - State University of New York, Syracuse, New York
  - University of Vermont Department of Neurology, Burlington, Vermont

REFERENCES:
- [Background] AAEM Quality Assurance Committee. American Association of Electrodiagnostic Medicine. Practice parameter for repetitive nerve stimulation and single fiber EMG evaluation of adults with suspected myasthenia gravis or Lambert-Eaton myasthenic syndrome: summary statement. Muscle Nerve. 2001 Sep;24(9):1236-8. doi: 10.1002/mus.1139. No abstract available. PMID 11494280
- [Background] Aranda JM Jr, Scornik JC, Normann SJ, Lottenberg R, Schofield RS, Pauly DF, Miles M, Hill JA, Sleasman JW, Skoda-Smith S. Anti-CD20 monoclonal antibody (rituximab) therapy for acute cardiac humoral rejection: a case report. Transplantation. 2002 Mar 27;73(6):907-10. doi: 10.1097/00007890-200203270-00013. PMID 11923690
- [Background] Barohn RJ, McIntire D, Herbelin L, Wolfe GI, Nations S, Bryan WW. Reliability testing of the quantitative myasthenia gravis score. Ann N Y Acad Sci. 1998 May 13;841:769-72. doi: 10.1111/j.1749-6632.1998.tb11015.x. No abstract available. PMID 9668327
- [Background] Besinger UA, Toyka KV, Homberg M, Heininger K, Hohlfeld R, Fateh-Moghadam A. Myasthenia gravis: long-term correlation of binding and bungarotoxin blocking antibodies against acetylcholine receptors with changes in disease severity. Neurology. 1983 Oct;33(10):1316-21. doi: 10.1212/wnl.33.10.1316. PMID 6684226
- [Background] Chemnitz J, Draube A, Scheid C, Staib P, Schulz A, Diehl V, Sohngen D. Successful treatment of severe thrombotic thrombocytopenic purpura with the monoclonal antibody rituximab. Am J Hematol. 2002 Oct;71(2):105-8. doi: 10.1002/ajh.10204. PMID 12353309
- [Background] Chiu HC, Chen WH, Yeh JH. The six year experience of plasmapheresis in patients with myasthenia gravis. Ther Apher. 2000 Aug;4(4):291-5. doi: 10.1046/j.1526-0968.2000.004004291.x. PMID 10975476
- [Background] Dallaire B, Leonard J, Varns C et al. IDEC-C2B8 (Rituximab): Biology and preclinical studies. J Mol Med 75:B230, 1997.
- [Background] Davis TA, Grillo-Lopez AJ, White CA, McLaughlin P, Czuczman MS, Link BK, Maloney DG, Weaver RL, Rosenberg J, Levy R. Rituximab anti-CD20 monoclonal antibody therapy in non-Hodgkin's lymphoma: safety and efficacy of re-treatment. J Clin Oncol. 2000 Sep;18(17):3135-43. doi: 10.1200/JCO.2000.18.17.3135. PMID 10963642
- [Background] Gajra A, Vajpayee N, Grethlein SJ. Response of myasthenia gravis to rituximab in a patient with non-Hodgkin lymphoma. Am J Hematol. 2004 Oct;77(2):196-7. doi: 10.1002/ajh.20169. PMID 15389902
- [Background] Grollo-Lopez A, Varns C, Waldichuk C et al. IDEC-C2B8 chimeric anti-CD20 antibody: Safety and clinical activity in the treatment of patients with relapsed low-grade or follicular (IWF:A-D) non-Hodgkin's lymphoma (NHL). Br J Haematol 93:283, 1996.
- [Background] Grob D. Natural history of myasthenia gravis. In: Engel AG (ed). Myasthenia Gravis and Myasthenic Disorders. New York: Oxford University Press, 1999, pp 131-145.
- [Background] Hilkevich O, Drory VE, Chapman J, Korczyn AD. The use of intravenous immunoglobulin as maintenance therapy in myasthenia gravis. Clin Neuropharmacol. 2001 May-Jun;24(3):173-6. doi: 10.1097/00002826-200105000-00010. PMID 11391130
- [Background] Jaretzki A 3rd, Barohn RJ, Ernstoff RM, Kaminski HJ, Keesey JC, Penn AS, Sanders DB. Myasthenia gravis: recommendations for clinical research standards. Task Force of the Medical Scientific Advisory Board of the Myasthenia Gravis Foundation of America. Neurology. 2000 Jul 12;55(1):16-23. doi: 10.1212/wnl.55.1.16. No abstract available. PMID 10891897
- [Background] Jenkins D, DiFrancesco L, Chaudhry A, Morris D, Gluck S, Jones A, Woodman R, Brown CB, Russell J, Stewart DA. Successful treatment of post-transplant lymphoproliferative disorder in autologous blood stem cell transplant recipients. Bone Marrow Transplant. 2002 Sep;30(5):321-6. doi: 10.1038/sj.bmt.1703603. PMID 12209355
- [Background] Leget GA, Czuczman MS. Use of rituximab, the new FDA-approved antibody. Curr Opin Oncol. 1998 Nov;10(6):548-51. doi: 10.1097/00001622-199811000-00012. PMID 9818234
- [Background] Levine TD, Pestronk A. IgM antibody-related polyneuropathies: B-cell depletion chemotherapy using Rituximab. Neurology. 1999 May 12;52(8):1701-4. doi: 10.1212/wnl.52.8.1701. PMID 10331706
- [Background] Mantegazza R, Antozzi C, Peluchetti D, Sghirlanzoni A, Cornelio F. Azathioprine as a single drug or in combination with steroids in the treatment of myasthenia gravis. J Neurol. 1988 Nov;235(8):449-53. doi: 10.1007/BF00314245. PMID 3062134
- [Background] Oosterhuis HJ. The natural course of myasthenia gravis: a long term follow up study. J Neurol Neurosurg Psychiatry. 1989 Oct;52(10):1121-7. doi: 10.1136/jnnp.52.10.1121. PMID 2795037
- [Background] Osserman KE, Genkins G. Studies in myasthenia gravis: review of a twenty-year experience in over 1200 patients. Mt Sinai J Med. 1971 Nov-Dec;38(6):497-537. No abstract available. PMID 4941403
- [Background] Pascuzzi RM, Coslett HB, Johns TR. Long-term corticosteroid treatment of myasthenia gravis: report of 116 patients. Ann Neurol. 1984 Mar;15(3):291-8. doi: 10.1002/ana.410150316. PMID 6721451
- [Background] Paul RH, Nash JM, Cohen RA, Gilchrist JM, Goldstein JM. Quality of life and well-being of patients with myasthenia gravis. Muscle Nerve. 2001 Apr;24(4):512-6. doi: 10.1002/mus.1034. PMID 11268023
- [Background] Reff ME, Carner K, Chambers KS, Chinn PC, Leonard JE, Raab R, Newman RA, Hanna N, Anderson DR. Depletion of B cells in vivo by a chimeric mouse human monoclonal antibody to CD20. Blood. 1994 Jan 15;83(2):435-45. PMID 7506951
- [Background] Seybold ME. Diagnosis of myasthenia gravis. In: Engel AG (ed). Myasthenia Gravis and Myasthenic Disorders. New York: Oxford University Press, 1999, pp 146-166.
- [Background] Seybold ME. Treatment of myasthenia gravis. In: Engel AG (ed). Myasthenia Gravis and Myasthenic Disorders. New York: Oxford University Press, 1999a, pp 167-201.
- [Background] Tindall RS, Phillips JT, Rollins JA, Wells L, Hall K. A clinical therapeutic trial of cyclosporine in myasthenia gravis. Ann N Y Acad Sci. 1993 Jun 21;681:539-51. doi: 10.1111/j.1749-6632.1993.tb22937.x. PMID 8357194
- [Background] Wolfe GI, Herbelin L, Nations SP, Foster B, Bryan WW, Barohn RJ. Myasthenia gravis activities of daily living profile. Neurology. 1999 Apr 22;52(7):1487-9. doi: 10.1212/wnl.52.7.1487. PMID 10227640
- [Background] Zaja F, Russo D, Fuga G, Perella G, Baccarani M. Rituximab for myasthenia gravis developing after bone marrow transplant. Neurology. 2000 Oct 10;55(7):1062-3. doi: 10.1212/wnl.55.7.1062-a. No abstract available. PMID 11061276
- [Background] Zecca M, De Stefano P, Nobili B, Locatelli F. Anti-CD20 monoclonal antibody for the treatment of severe, immune-mediated, pure red cell aplasia and hemolytic anemia. Blood. 2001 Jun 15;97(12):3995-7. doi: 10.1182/blood.v97.12.3995. PMID 11389047